CLINICAL TRIAL: NCT00109876
Title: A Pilot Study of Radiofrequency Ablation in High-Risk Patients With Stage IA Non-Small Cell Lung Cancer
Brief Title: Radiofrequency Ablation in Treating Patients With Stage I Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z4033; ACOSOG-Z4033; CDR0000426417 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RFA therapy) (Experimental): A radiofrequency electrode is placed by CT guidance into the target tumor. Patients undergo RFA directly to the tumor for up to 12 minutes to obtain an intratumoral temperature > 60° C. Patients may receive 3 RFA treatments (a total of 36 minutes) to obtain the target temperature.
  Interventions: Procedure: Computed Tomography-Guided Optical Sensor-Guided Radiofrequency Ablation

INTERVENTIONS:
Procedure: Computed Tomography-Guided Optical Sensor-Guided Radiofrequency Ablation — Undergo RFA
  Other Names: CT-guided optical sensor-guided radiofrequency ablation, CT-guided optical sensor-guided RF ablation

SUMMARY:
This pilot clinical trial studies how well radiofrequency ablation works in treating patients with stage IA non-small cell lung cancer. Radiofrequency ablation uses high-frequency electric current to kill tumor cells. Computed tomography (CT)-guided radiofrequency ablation may be a better treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the overall 2-year survival rate after radiofrequency ablation (RFA).

SECONDARY OBJECTIVES:

I. To assess freedom from regional or distant recurrence. II. To assess freedom from local recurrence in the ablated lobe. III. To estimate the number of procedures deemed technical successes. IV. To evaluate procedure-specific morbidity and mortality. V. To explore the utility of immediate (within 96 hours) post-RFA positron emission tomography (PET) in predicting overall survival and local control.

VI. To explore the effect of RFA on both short-term (3 months post-RFA) and long-term (24 months post-RFA) pulmonary function.

OUTLINE:

A radiofrequency electrode is placed by CT guidance into the target tumor. Patients undergo RFA directly to the tumor for up to 12 minutes to obtain an intratumoral temperature > 60° Celsius (C). Patients may receive 3 RFA treatments (a total of 36 minutes) to obtain the target temperature.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION CRITERIA:
* Patients must have a lung nodule suspicious for clinical stage I non-small cell lung cancer (NSCLC)
* Patient must have a mass =< 3 cm maximum diameter by CT size estimate: clinical stage IA
* Patient must have been evaluated by a thoracic surgeon and been deemed at high risk for a lung resection; NOTE: if the evaluating surgeon is not a member of American College of Surgeons Oncology Group (ACOSOG), then an ACOSOG thoracic surgeon must confirm with dated signature that the patient is high-risk and appropriate for RFA
* Patient must have fludeoxyglucose F 18 (FDG)-PET and a CT scan of the chest with upper abdomen within 60 days prior to pre-registration; patient must have pulmonary function tests (PFTs) within 120 days prior to registration
* Patient must have an Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status 0, 1, or 2
* Patient must meet at least one major criterion or meet a minimum of two minor criteria as described below:

  * Major criteria

    * Forced expiratory volume in one second (FEV1) =< 50% predicted
    * Diffusing capacity of the lung for carbon monoxide (DLCO) =< 50% predicted
  * Minor Criteria

    * Age >= 75
    * FEV1 51-60% predicted
    * DLCO 51-60% predicted
    * Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40 mmHg) as estimated by echocardiography or right heart catheterization
    * Poor left ventricular function (defined as an ejection fraction of 40% or less)
    * Resting or exercise arterial partial pressure of oxygen (pO2) =< 55 mmHg or oxygen saturation (SpO2) =< 88%
    * Partial pressure of carbon dioxide (pCO2) > 45 mmHg
    * Modified Medical Research Council (MMRC) Dyspnea Scale >= 3
* Patient must not have had previous intra-thoracic radiation therapy
* Women of child-bearing potential must have negative serum or urine pregnancy test within 2 weeks of registration
* REGISTRATION ACTIVATION CRITERIA:
* Patient must have histologically or cytologically proven NSCLC, 3 cm or smaller, as determined by the largest dimension on CT lung windows
* Patient's tumor must be non-contiguous with vital structures: trachea, esophagus, aorta, aortic arch branches and heart and lesions must be accessible via percutaneous transthoracic route
* Patient must have all suspicious mediastinal lymph nodes (> 1 cm short-axis dimension on CT scan or positive on PET scan) assessed by the following to confirm negative involvement with NSCLC (mediastinoscopy, endo-esophageal ultrasound-guided needle aspiration, CT-guided, video-assisted thoracoscopic or open lymph node biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-09; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damian E. Dupuy, MD, Study Chair — Rhode Island Hospital
Locations (17):
- United States (17):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Good Samaritan Hospital Cancer Treatment Center, Cincinnati, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - H. Clay Evans Johnson Cancer Center at Memorial Hospital, Chattanooga, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-four (54) participants were enrolled from 16 institutions from December 2006 to November 2010.
Pre-assignment Details: Two participants had pre-RFA positron emission tomography (PET) not within 60 days before study preregistration and one participant did not had non-small cell lung cancer, which were deemed ineligible for the studies, and were excluded from all analyses.
Groups:
- RFA Therapy: Patients undergo radiofrequency ablation (RFA) directly to the tumor for up to 12 minutes to obtain an intratumoral temperature > 60° C. Patients may receive 3 RFA treatments (a total of 36 minutes) to obtain the target temperature.
Period: Overall Study
Arm/Group | RFA Therapy
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who met the eligibility criteria.
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 76 [60 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 51
Eastern Cooperative Oncology Group (ECOG)Performance Status [Count of Participants; unit: Participants]
  0 = Asymptomatic and fully active | 9
  1= Symptomatic and fully ambulatory | 29
  2= Symptomatic and ambulatory | 13
Baseline Forced Expiratory Volume in 1 second (FEV1) [Median (Full Range); unit: Percentage of predicted] | 48 [13 to 102]
Baseline diffusing capacity of the lung for carbon monoxide (DLCO) [Median (Full Range); unit: Percentage of predicted] | 42 [7 to 99]
Baseline forced vital capacity [Median (Full Range); unit: mL] | 2070 [1090 to 3720]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 2 Years
Description: Percentage of participants who were alive at 2 years. The 2 year survival was estimated using the Kaplan Meier method.
Time Frame: 2 years from registration
Population: All enrolled participants who met the eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
percentage of participants | 69.8 [58.0 to 83.9]

2. Secondary Outcome: Overall Time to Local Failure
Description: The overall time to local failure was defined as the time from registration to documentation of > local failure. The local failure was defined as the recurrence in the same lobe or hilum (N1 nodes) or progression at the ablated site after treatment affects have subsided.
Time Frame: Up to 2 years
Population: All enrolled participants who met the eligibility criteria.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
years | NA [1.17 to NA] — The median of time to local failure and upper limit of 95% confidence interval are not attainable.

3. Secondary Outcome: Overall Time to Recurrence
Description: The overall time to recurrence was defined as the time from registration to documentation of disease recurrence. If a patient dies without a documentation of disease recurrence, the patient will be considered to have had tumor recurrence at the time of their death unless there is sufficient evidence to conclude no recurrence occurred prior to death.
Time Frame: Up to 2 years
Population: All enrolled participants who met the eligibility criteria.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
years | 1.40 [0.75 to NA] — The upper limit of 95% confidence interval is not attainable.

4. Secondary Outcome: Number of Procedures Deemed Technical Successes
Description: The number of procedures deemed technical successes is defined as the number of patients with a RFA procedures deemed a technical success. A technical success is defined as follows: The pertinent captured images from the treatment CT showing RFA electrode placement and the recorded RFA generator parameters (e.g. impedance, current, power, treatment time and maximum intra-tumoral temperature) were reviewed by the quality control panel to determine technical success.
Time Frame: Up to 2 years
Population: All enrolled participants who met the eligibility criteria.
Measure: Number; unit: number of technical successes
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
number of technical successes | 50

5. Secondary Outcome: Incidence of Adverse Events
Description: The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 was used to evaluate adverse event.> Grade 1: mild; Grade 2: moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death.
Time Frame: Up to 2 years
Population: All enrolled participants who met the eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
Participants
  Grade 0 Adverse Events | 22
  Grade 1 Adverse Events | 5
  Grade 2 Adverse Events | 6
  Grade 3 Adverse Events | 12
  Grade 4 Adverse Events | 3
  Grade 5 Adverse Events | 3

6. Secondary Outcome: Change in Pulmonary Function From Baseline at Month 3
Description: Pulmonary function test values include forced expiratory volume 1 (FEV1) and carbon monoxide diffusion (DLCO). The distribution of clinically meaningful changes (10% increase or 10% decrease) in pulmonary function from the baseline to 3 was summarized.
Time Frame: Baseline and Month 3
Population: All enrolled participants who met the eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
Participants
  FEV1, % predicted: Missing | 12
  FEV1, % predicted: 10% increase | 5
  FEV1, % predicted: 10% decrease | 3
  FEV1, % predicted: Neither increase nor decrease of 10% | 31
  DLCO, % predicted: Missing | 17
  DLCO, % predicted: 10% increase | 9
  DLCO, % predicted: 10% decrease | 4
  DLCO, % predicted: Neither increase nor decrease of 10% | 21

7. Secondary Outcome: Change in Pulmonary Function From Baseline at Month 24
Description: Pulmonary function test values include forced expiratory volume 1 (FEV1) and carbon monoxide diffusion (DLCO). The distribution of clinically meaningful changes (10% increase or 10% decrease) in pulmonary function from the baseline to 24 was summarized.
Time Frame: Baseline and Month 24
Population: All enrolled participants who met the eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | RFA Therapy
Number analyzed (Participants) | 51
Participants
  FEV1, % predicted: Missing | 30
  FEV1, % predicted: 10% increase | 7
  FEV1, % predicted: 10% decrease | 4
  FEV1, % predicted: Neither increase nor decrease of 10% | 10
  DLCO, % predicted: Missing | 35
  DLCO, % predicted: 10% increase | 6
  DLCO, % predicted: 10% decrease | 4
  DLCO, % predicted: Neither increase nor decrease of 10% | 6

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events are described and graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 3.0.
Arm/Group | RFA Therapy
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 29/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RFA Therapy (N=51)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 4 (4)
Cardiac troponin I increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less